CLINICAL TRIAL: NCT05809271
Title: Acute Effects of 3,4-methylenedioxymethamphetamine (MDMA) With and Without a Booster Dose (MDMA-booster Study)
Brief Title: Acute Effects of 3,4-methylenedioxymethamphetamine (MDMA) With and Without a Booster Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2023-00167
Record Dates: First submitted 2023-03-13; First posted 2023-04-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: 3-period, random order, placebo-controlled, double-blind cross-over study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MDMA with booster (Experimental): MDMA followed by MDMA
  Interventions: Drug: MDMA 120 mg + MDMA 60 mg
- MDMA without booster (Experimental): MDMA followed by placebo
  Interventions: Drug: MDMA 120 mg + placebo
- Placebo (Placebo Comparator): Placebo followed by placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDMA 120 mg + MDMA 60 mg — An oral dose of 120 mg racemic MDMA will be administered followed by a second dose of 60 mg racemic MDMA two hours later.
  Other Names: 3,4-Methylenedioxymethamphetamine
  Arms: MDMA with booster
Drug: MDMA 120 mg + placebo — An oral dose of 120 mg racemic MDMA will be administered followed by a placebo two hours later.
  Other Names: 3,4-Methylenedioxymethamphetamine
  Arms: MDMA without booster
Drug: Placebo — An oral placebo will be administered followed by a placebo two hours later.
  Arms: Placebo

SUMMARY:
3,4-methylenedioxymethamphetamine (MDMA) is a psychoactive substance and prototypical empathogen acutely inducing feelings of heightened mood, empathy, trust and closeness to others. The current study investigates differences in duration of acute effects and side effects after administration of a single dose of MDMA compared to a repeated administration.

DETAILED DESCRIPTION:
MDMA is a psychoactive substance that primarily enhances serotonergic neurotransmission by releasing 5-HT through the SERT. It also releases dopamine and norepinephrine, although less potently, through the dopamine transporter and norepinephrine transporter, respectively. In addition to its use as a recreational drug, MDMA-assisted psychotherapy has been investigated in several phase 2 trials and one phase 3 trial for PTSD. Further indications for MDMA-assisted therapy being planned or ongoing are eating disorders, social anxiety, and alcohol use disorder.

The present study focuses on dosing aspects of MDMA used in clinical studies and recreational settings, specifically the benefits of a second administration (booster dose) given several hours after the initial dose. Most published studies of MDMA-assisted psychotherapy used a booster dose. A typical dosing regimen would be 80-120 mg of MDMA initially followed by half the initial dose after 1.5-2.5 hours. Although previous studies have found that a booster dose could prolong the acute effects of MDMA, others have shown an acute tolerance reflected in the finding that acute subjective effects return to baseline within 4-5 hours, while plasma concentrations are still close to peak levels.

These findings have led to controversy regarding how effective a booster dose would be in prolonging acute effects, as it has never been directly compared to placebo. Additionally, the higher total dose could lead to an increase in side effects.

Therefore, the present phase 1 study intends to compare the acute subjective, physiological, and endocrine effects of MDMA (120 mg + 60 mg after 2 hours), MDMA (120 mg + placebo after 2 hours), and (placebo + placebo after 2 hours) using a double-blind, random-order, crossover design in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Good understanding of the German language.
2. Understanding the procedures and the risks that are associated with the study.
3. Participants must be willing to adhere to the protocol and sign the consent form.
4. Participants must be willing to refrain from taking illicit psychoactive substances during the study.
5. Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drinks after midnight of the evening before the study session, as well as during the study day.
6. Participants must be willing not to drive a traffic vehicle or to operate machines within 48h after substance administration.
7. Willing to use effective birth control throughout study participation.
8. Body mass index between 18-29 kg/m2.

Exclusion Criteria:

1. Relevant chronic or acute medical condition.
2. Current or previous major psychiatric disorder.
3. Psychotic disorder in first-degree relatives, not including psychotic disorders secondary to an apparent medical reason, e.g. brain injury, dementia, or lesions of the brain.
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg).
5. Previous MDMA use more than 20 times or any time within the previous month.
6. Pregnant or nursing women.
7. Participation in another clinical trial (currently or within the last 30 days).
8. Use of medications that may interfere with the effects of the study medications.
9. Tobacco smoking (>10 cigarettes/day).
10. Consumption of alcoholic drinks (>15 drinks/week).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Subjective effect duration for "any drug effect" | Every 15 minutes for 9 hours after substance administration
  Assessed by visual analog scale (VAS) using 10% of the individual maximal subjective response (Emax) as threshold for the onset and offset.

SECONDARY OUTCOMES:
Maximal subjective effects for "any drug effect" | Every 15 minutes for 9 hours after substance administration
  Maximal subjective response (Emax), of "any drug effect" assessed by visual analog scale (VAS).
Total subjective effects for "any drug effect" | Every 15 minutes for 9 hours after substance administration
  Area under the effect curve (AUEC) of "any drug effect" assessed by visual analog scale (VAS).
Further acute subjective effects I duration | Every 30 minutes for 9 hours after substance administration
  Effect duration for "good drug effect", "bad drug effect", "liking", "stimulated", "high", "anxiety", "I am emotional", "talkative", "happy", "open", "trust", "feeling close to others", "want to be alone", and "want to be with others", assessed by visual analog scale (VAS) using 10% of the individual maximal subjective response (Emax) as threshold for the onset and offset.
Further acute subjective effects II maximal effects | Every 30 minutes for 9 hours after substance administration
  Maximal subjective response (Emax) of "good drug effect", "bad drug effect", "liking", "stimulated", "high", "anxiety", "I am emotional", "talkative", "happy", "open", "trust", "feeling close to others", "want to be alone", and "want to be with others", assessed by visual analog scale (VAS).
Further acute subjective effects III total effects | Every 30 minutes for 9 hours after substance administration
  Area under the effect curve (AUEC) of "good drug effect", "bad drug effect", "liking", "stimulated", "high", "anxiety", "I am emotional", "talkative", "happy", "open", "trust", "feeling close to others", "want to be alone", and "want to be with others", assessed by visual analog scale (VAS).
Further acute subjective effects IV AMRS | 5 times during each study day: 30 minutes before as well as 2, 4, 6, and 9 hours after substance administration.
  The Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely".
Acute autonomic effects I (blood pressure) | 16 times during each study day: 30 minutes before as well as 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9 hours after substance administration
  Blood pressure (systolic and diastolic) will be measured with an automatic oscillometric device.
Acute autonomic effects II (heart rate) | 16 times during each study day: 30 minutes before as well as 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9 hours after substance administration
  Heart rate will be measured with an automatic oscillometric device.
Acute autonomic effects III (body temperature) | 16 times during each study day: 30 minutes before as well as 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9 hours after substance administration
  Body temperature will be measured with an ear thermometer.
Adverse effects (acute and subacute) | Before each study day as baseline as well as 9 hours, 3 days and 7 days after substance administration
  The 2011 revised Beschwerden-Liste (B-LR) consists of a 40-item list covering a wide variety of symptoms and complaints that are answered with a four-point intensity-scoring ranging from "not at all" to "strong".
Subacute effects on general and mental well-being I (WEMWBS) | Before each study day as baseline as well as 3 days and 7 days after substance administration
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-item questionnaire, that covers different concepts associated with positive mental health, including both hedonic and eudaimonic aspects, positive affect, satisfying interpersonal relationships and positive functioning. For each item an ordinal five-point frequency answer format, ranging from 1 = none of the time" to 5 = "all of the time" is applied.
Subacute effects on general and mental well-being II (GHQ-12) | Before each study day as baseline as well as 3 days and 7 days after substance administration
  The General Health Questionnaire (GHQ-12) consists of a 12-item questionnaire with a four-point response scale assessing general psychological discomfort.
Subacute effects on general and mental well-being III (SPANE) | Before each study day as baseline as well as 3 days and 7 days after substance administration
  The Scale of Positive and Negative Experience (SPANE) is a 12-item questionnaire to capture the affective component of subjective well-being. The SPANE includes six items to assess positive feelings and six items to assess negative feelings. The feelings are reported on a 5-point scale ranging from "very rarely" to "very often or always".
Subacute effects on subjective sleep quality (ISI) | Before each study day as baseline as well as 3 days and 7 days after substance administration
  The Insomnia Severity Index (ISI) is a self-report instrument to assess subjective sleep complaints, screen for insomnia and evaluate treatment response. It consists of seven items scored on a five-point Likert-scale.
Plasma concentrations of MDMA | 16 times during each study day: 30 minutes before as well as 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9 hours after substance administration
  Assessed via blood samples. Findings will be described descriptively including maximal concentration (Cmax), time to Cmax, (Tmax) area under the concentration-time curve up to 9 h (AUC0-9) and elimination half-life values.
Plasma concentrations of MDMA-metabolites | 16 times during each study day: 30 minutes before as well as 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9 hours after substance administration
  Assessed via blood samples. Findings will be described descriptively including maximal concentration (Cmax), time to Cmax, (Tmax) area under the concentration-time curve up to 9 h (AUC0-9) and elimination half-life values.
Plasma concentrations of Plasma levels of oxytocin | 4 times during each study day: 30 minutes before as well as 2, 4 and 6 hours after substance administration
  Assessed via blood samples.
Effects on life satisfaction, well-being and appreciation before and after study I (BFW/E) | Twice during study: at screening and at end of study 12-14 weeks later.
  The "Positive Attitude towards Life" is an 8-item subscale of the 39-item Bern Subjective Well-Being Questionnaire for Adolescents (BFW/E). The BFW enables a reliable and valid assessment of different dimensions of subjective well-being in adolescents and adults. Changes over the course of the study are assessed.
Effects on life satisfaction, well-being and appreciation before and after study II (GLS) | Twice during study: at screening and at end of study 12-14 weeks later.
  Global life satisfaction is assessed based on a single item life satisfaction measure. The question can be answered on a 11-point scale: "In general, how satisfied are you with your life if 0 means 'not at all satisfied' and 10 means 'completely satisfied'?". Changes over the course of the study are assessed.
Effect moderation by personality traits I (NEO-FFI) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The NEO Five Factor Inventory (NEO-FFI) is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Effect moderation by personality traits II (FPI-R) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Freiburger Personality Inventory (FPI-R) version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Effect moderation by personality traits III (SPF) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Saarbrücker Persönlichkeitsfragebogen (SPF) defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
Effect moderation by personality traits IV (HEXACO) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The HEXACO personality inventory is a six-dimensional model of human personality with 100 items.The six factors are: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness and Openness to Experience.
Effect moderation by personality traits V (DSQ-40) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Defense Style Questionnaire (DSQ-40) can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Prof. Dr. MD, Principal Investigator — University Hospital Basel, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland